CLINICAL TRIAL: NCT02142517
Title: Comparative Study Between Duct to Mucosa and Invagination Pancreaticojejunostomy After Pancreaticoduodenectomy: A Prospective Randomized Study
Brief Title: Comparative Study Between Duct to Mucosa and Invagination Pancreaticojejunostomy After Pancreaticoduodenectomy:
Acronym: PJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, Ass. Prof., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pancreatic reconstruction
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2011-06

CONDITIONS: Pancreatic Anastomotic Leak
Keywords: pancreaticoduodenectomy, pancreatic fistula
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duct to mucosa PJ group (Active Comparator): Duct to mucosa PJ was performed by a two layer end to side PJ. The pancreatic capsule and jejunal serosa were anastomosed by interrupted silk suture 3/0 to form the outer layer in both the anterior and posterior wall of the anastomosis. Jejunostomy was done matched to the pancreatic duct diameter. The inner layer duct to mucosa was performed in eight to twelve stitches with 5/0 prolene. A pancreatic duct stent was inserted during anastomosis to allow easy and accurate suture placement, ensure adequate pancreatic duct exposure, and protect the opposite wall from being inadvertently held by needles then it was removed at the end of anastomosis.
  Interventions: Procedure: Duct to mucosa PJ group
- Invagination PJ group (Active Comparator): Invagination PJ was performed as an end to side. The pancreatic capsule and jejunal serosa were anastomosed by interrupted silk suture 3/0 to form the outer layer in both the anterior and posterior wall of the anastomosis. Jejunostomy was done matched to the pancreatic stump diameter. The inner layer was performed with 5/0 prolene between pancreatic parenchyma and mucosa. The duct was taken posteriorly and anteriorly to jejunal mucosa. A pancreatic duct stent was inserted during anastomosis and removed at the end of taking the stitches. Reconstruction was completed by end to side hepaticojejunostomy (retrocolic) and gastrojejunostomy (GJ) (antecolic) end to side manually.
  Interventions: Procedure: Invagination PJ group

INTERVENTIONS:
Procedure: Duct to mucosa PJ group — Duct to mucosa PJ was performed by a two layer end to side PJ. The pancreatic capsule and jejunal serosa were anastomosed by interrupted silk suture 3/0 to form the outer layer in both the anterior and posterior wall of the anastomosis. Jejunostomy was done matched to the pancreatic duct diameter. The inner layer duct to mucosa was performed in eight to twelve stitches with 5/0 prolene. A pancreatic duct stent was inserted during anastomosis to allow easy and accurate suture placement, ensure adequate pancreatic duct exposure, and protect the opposite wall from being inadvertently held by needles then it was removed at the end of anastomosis.
  Other Names: Group 1
  Arms: Duct to mucosa PJ group
Procedure: Invagination PJ group — Invagination PJ was performed as an end to side. The pancreatic capsule and jejunal serosa were anastomosed by interrupted silk suture 3/0 to form the outer layer in both the anterior and posterior wall of the anastomosis. Jejunostomy was done matched to the pancreatic stump diameter. The inner layer was performed with 5/0 prolene between pancreatic parenchyma and mucosa. The duct was taken posteriorly and anteriorly to jejunal mucosa. A pancreatic duct stent was inserted during anastomosis and removed at the end of taking the stitches. Reconstruction was completed by end to side hepaticojejunostomy (retrocolic) and gastrojejunostomy (GJ) (antecolic) end to side manually.
  Other Names: Group 2
  Arms: Invagination PJ group

SUMMARY:
Postoperative pancreatic fistula (POPF) remains a challenge even at specialized centers, and also affect significantly the surgical outcomes . The incidence of POPF after pancreaticoduodenectomy among different studies, ranging from 5 to 30%.Morbidity and mortality after pancreaticoduodenectomy are usually related to surgical management of the pancreatic stump. The safe pancreatic reconstruction after pancreaticoduodenectomy continues to be a challenge at high volume centers. The variety of reconstruction is a reflection of the lack of ideal one.Duct to mucosa and invagination are two classic PJ techniques. Many studies compared both techniques, but their surgical outcomes still unclear.The aim of the study was to assess the effectiveness and surgical outcomes of both techniques of PJ after pancreaticoduodenectomy.

DETAILED DESCRIPTION:
Consecutive patients who were treated by pancreaticoduodenectomy at Gastroenterology Surgical Center, Mansoura, Egypt Exclusion criteria included any patients with locally advanced periampullary tumour, metastases, patients received neoadjuvant chemoradiotherapy, patients underwent pancreaticogastrostomy (PG), patients with advanced liver cirrhosis (Child B or C), malnutrition, or coagulopathy.

All patients were subjected to careful history taking, clinical examination, routine laboratory investigation abdominal ultrasound, magnetic resonance cholangiopancreatography , and abdominal computerized tomography .

The patients were randomized into two groups: Group I: patients underwent duct to mucosa PJ. Group II: patients underwent invagination PJ.

The primary outcome was POPF rate.Secondary outcomes were operative time, operative time needed for reconstruction, length of postoperative hospital stay, postoperative morbidities

ELIGIBILITY:
Inclusion Criteria:

-Consecutive patients who were treated by pancreaticoduodenectomy

Exclusion Criteria:

* Any patients with locally advanced periampullary tumour, metastases
* Patients received neoadjuvant chemoradiotherapy
* Patients underwent pancreaticogastrostomy (PG)
* Patients with advanced liver cirrhosis (Child B or C)
* Malnutrition
* Coagulopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
POPF | up to 30 days
  POPF was defined by International Study Group of Pancreatic Fistula (ISGPF) as any measurable volume of fluid on or after POD 3 with amylase content greater than 3 times the serum amylase activity . A pancreatic fistula (PF) were graded according to the ISGPF into Grade A, B, and C according to the clinical course

SECONDARY OUTCOMES:
operative time | up to 10 hours
  time of surgical procedure
hospital stay | up to 60 days
  postoperative stay
postoperative complications | up to 90 days
  delayed gastric emptying (DGE), pancreatitis, biliary leakage
Pancreatic function | up to one year
  Pancreatic exocrine function was evaluated clinically. It was assessed by presence or absence of steatorrhae (more than three stool per day, fecal output of > 200 g/d for at least three days, pale or yellow stools, and appearance of stools as pasty or greasy, the need of pancreatic enzymes supplement and studied variation in body weight pre and postoperative (

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El Nakeeb, MD, Principal Investigator — Mansoura University
Locations (1):
- Ayman El Nakeeb, Al Mansurah, Mansoura, Egypt

REFERENCES:
- [Result] El Nakeeb A, Salah T, Sultan A, El Hemaly M, Askr W, Ezzat H, Hamdy E, Atef E, El Hanafy E, El-Geidie A, Abdel Wahab M, Abdallah T. Pancreatic anastomotic leakage after pancreaticoduodenectomy. Risk factors, clinical predictors, and management (single center experience). World J Surg. 2013 Jun;37(6):1405-18. doi: 10.1007/s00268-013-1998-5. PMID 23494109
- [Result] Bassi C, Falconi M, Molinari E, Mantovani W, Butturini G, Gumbs AA, Salvia R, Pederzoli P. Duct-to-mucosa versus end-to-side pancreaticojejunostomy reconstruction after pancreaticoduodenectomy: results of a prospective randomized trial. Surgery. 2003 Nov;134(5):766-71. doi: 10.1016/s0039-6060(03)00345-3. PMID 14639354
- [Result] Hayashibe A, Kameyama M. The clinical results of duct-to-mucosa pancreaticojejunostomy after pancreaticoduodenectomy in consecutive 55 cases. Pancreas. 2007 Oct;35(3):273-5. doi: 10.1097/MPA.0b013e3180676dc2. PMID 17895850
- [Result] Hosotani R, Doi R, Imamura M. Duct-to-mucosa pancreaticojejunostomy reduces the risk of pancreatic leakage after pancreatoduodenectomy. World J Surg. 2002 Jan;26(1):99-104. doi: 10.1007/s00268-001-0188-z. Epub 2001 Nov 26. PMID 11898041
- [Result] Zhang JL, Xiao ZY, Lai DM, Sun J, He CC, Zhang YF, Chen S, Wang J. Comparison of duct-to-mucosa and end-to-side pancreaticojejunostomy reconstruction following pancreaticoduodenectomy. Hepatogastroenterology. 2013 Jan-Feb;60(121):176-9. doi: 10.5754/hge12496. PMID 22773303
- [Result] Bai XL, Zhang Q, Masood N, Masood W, Gao SL, Zhang Y, Shahed S, Liang TB. Duct-to-mucosa versus invagination pancreaticojejunostomy after pancreaticoduodenectomy: a meta-analysis. Chin Med J (Engl). 2013 Nov;126(22):4340-7. PMID 24238526
- [Derived] El Nakeeb A, El Hemaly M, Askr W, Abd Ellatif M, Hamed H, Elghawalby A, Attia M, Abdallah T, Abd ElWahab M. Comparative study between duct to mucosa and invagination pancreaticojejunostomy after pancreaticoduodenectomy: a prospective randomized study. Int J Surg. 2015 Apr;16(Pt A):1-6. doi: 10.1016/j.ijsu.2015.02.002. Epub 2015 Feb 13. PMID 25682724
- See also: Mansoura university, Mansoura, Egypt — http://www.mans.edu.eg/